CLINICAL TRIAL: NCT06533488
Title: Evaluation of the Impact of a Perceptual Learning Module (PLM) on the Sonographic Identification of Spinal Structures by Novice Anesthesiology Residents. A Randomized Controlled Study
Brief Title: Evaluation of a Perceptual Learning Module on Spinal Ultrasound Among Residents.
Acronym: MAP-Rachis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Issam TANOUBI, MD, MA (Ed), DESAR, Maisonneuve-Rosemont Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2024-3447
Record Dates: First submitted 2024-04-02; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Spinal Anesthesia Skill; Ultrasound Imaging of Anatomical Structures; Medical Education

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Feedback group (Experimental): This group will receive feedback upon completion of the task.
  Interventions: Other: Perceptual learning module
- Control group (Placebo Comparator): This group will not receive any feedback
  Interventions: Other: Control

INTERVENTIONS:
Other: Perceptual learning module — Perceptual learning module providing feedback on the most relevant image for clinical practice in a spinal ultrasound video.
  Arms: Feedback group
Other: Control — Participants in the control group will view the same videos as participants in the intervention group without feedback on the best image.
  Arms: Control group

SUMMARY:
This medical education research project aims to evaluate the impact of a directed perceptual learning module (PLM) on spinal sonoanatomy. Following a demographic questionnaire, participants will be exposed to a tutorial explaining the necessary theoretical foundations for the PLM as well as the functioning of the PLM interface. A pre-test involving selecting the best image from a video sequence depicting spinal sonoanatomy will be administered to all participants. Participants will then be randomized into two groups and exposed to video sequences in the same manner as during the pre-test, with immediate feedback in the intervention group and no feedback in the control group. The video sequences presented will be the same between the two groups. Finally, a post-test will be administered immediately and remotely after exposure to the PLM. The time window corresponding to the best image will be predefined by an expert and compared to the resident's value. The difference in feedback exposure between the two groups will not be revealed to limit biases.

ELIGIBILITY:
Inclusion Criteria (participants) :

* To be a first, second, third, or fourth-year resident in the anesthesiology program at the Université de Montréal.
* Not having experience in spinal ultrasound (defined as not having performed more than 5 spinal ultrasounds, whether accompanied or not).
* To be familiar with ultrasound.
* Consenting to participate in the study.

Inclusion Criteria (experts) :

- Having used spinal ultrasound in clinical practice or taught it within the last year.

Exclusion Criteria (participants) :

* Refusal to consent
* Not meeting the inclusion criteria.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Improvement in the concordance of identifying the best image on the video within the interval specified by the expert in seconds, between the pre-test and the post-test. | Between the pre-test and the immediate post-test, as well as the post-test at 1 month.

SECONDARY OUTCOMES:
Improvement over time in the concordance of identifying the best image on the video within the interval specified by the expert in seconds | During the intervention phase

CONTACTS AND LOCATIONS:
Locations (1):
- Maisonneuve-Rosemont Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Guegan S, Steichen O, Soria A. Literature review of perceptual learning modules in medical education: What can we conclude regarding dermatology? Ann Dermatol Venereol. 2021 Mar;148(1):16-22. doi: 10.1016/j.annder.2020.01.023. Epub 2020 Jul 9. PMID 32654795
- [Result] Kellman PJ, Krasne S. Accelerating expertise: Perceptual and adaptive learning technology in medical learning. Med Teach. 2018 Aug;40(8):797-802. doi: 10.1080/0142159X.2018.1484897. Epub 2018 Aug 9. PMID 30091650
- [Result] VanderWielen BA, Harris R, Galgon RE, VanderWielen LM, Schroeder KM. Teaching sonoanatomy to anesthesia faculty and residents: utility of hands-on gel phantom and instructional video training models. J Clin Anesth. 2015 May;27(3):188-94. doi: 10.1016/j.jclinane.2014.07.007. Epub 2014 Nov 27. PMID 25433727
- [Result] Deacon AJ, Melhuishi NS, Terblanche NC. CUSUM method for construction of trainee spinal ultrasound learning curves following standardised teaching. Anaesth Intensive Care. 2014 Jul;42(4):480-6. doi: 10.1177/0310057X1404200409. PMID 24967763
- [Result] Watson MJ, Evans S, Thorp JM. Could ultrasonography be used by an anaesthetist to identify a specified lumbar interspace before spinal anaesthesia? Br J Anaesth. 2003 Apr;90(4):509-11. doi: 10.1093/bja/aeg096. PMID 12644427
- [Result] Ramlogan R, Niazi AU, Jin R, Johnson J, Chan VW, Perlas A. A Virtual Reality Simulation Model of Spinal Ultrasound: Role in Teaching Spinal Sonoanatomy. Reg Anesth Pain Med. 2017 Mar/Apr;42(2):217-222. doi: 10.1097/AAP.0000000000000537. PMID 28045758
- [Result] Chin KJ, Perlas A. Ultrasonography of the lumbar spine for neuraxial and lumbar plexus blocks. Curr Opin Anaesthesiol. 2011 Oct;24(5):567-72. doi: 10.1097/ACO.0b013e32834aa234. PMID 21822134
- [Result] Margarido CB, Arzola C, Balki M, Carvalho JC. Anesthesiologists' learning curves for ultrasound assessment of the lumbar spine. Can J Anaesth. 2010 Feb;57(2):120-6. doi: 10.1007/s12630-009-9219-2. Epub 2009 Dec 30. PMID 20041358
- [Result] Sidiropoulou T, Christodoulaki K, Siristatidis C. Pre-Procedural Lumbar Neuraxial Ultrasound-A Systematic Review of Randomized Controlled Trials and Meta-Analysis. Healthcare (Basel). 2021 Apr 17;9(4):479. doi: 10.3390/healthcare9040479. PMID 33920621